CLINICAL TRIAL: NCT06407895
Title: Effects of Lower Limb Fitness Program in Children With Down Syndrome
Brief Title: Effects of Lower Limb Fitness Program in Children With DS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: REC/RCR&AHS/23/0786
Record Dates: First submitted 2024-05-06; First posted 2024-05-09 (Actual); Last update posted 2024-08-02 (Actual); Status verified 2024-07

CONDITIONS: Down Syndrome
Keywords: Down Syndrome; Dynamic Balance; Lower Limb Fitness Program,
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Intervention Model Description: t will be Randomized control trial in which non probabilty convenient sampling will be used. Two groups of 6-10 age will be formed in which participants will be randomly divided. Group A will only receive Lower Limb Fitness Program and group B will receive Routine Therapy
Who Masked: Participant
Masking Description: Participants will get separate treatment protocols and possible efforts will be put to mask the both group about the treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lower Limb Fitness Program (Experimental): Group A will receive Range of motion for 5 minutes involving movements that stretch and strengthen the muscles and improve the stability. Proprioceptive training for 5 minutes which involve Single-leg balance Start with 20-30 seconds per leg and gradually increase to 1 minute 2-3 sets per leg. Weight bearing exercises on an uneven surface (such as Bosu ball or stability disc) and jumping rope 5-10 minutes/session. All proprioceptive training done firstly with eyes open and then with close eyes. Squat-to-stand training proprioceptive training lower extremity.
  Interventions: Other: Lower Limb Fitness Program
- Routine Therapy (Active Comparator): In control group routine therapy will be given 3 times a week for 6 weeks with session conducting 45 minutes per sessions which involve standing balance exercises, sitting from chair to stand, heal to toe stand will be performed.
  Interventions: Other: Routine Therapy

INTERVENTIONS:
Other: Lower Limb Fitness Program — the stability of the core area can help to improve dynamic balance, coordinate the upper and lower trunk muscles, and reduce muscles' damage and abnormalities. Physiotherapy had a role in programming training for Down Syndrome children, for example, using squat to stand training that seemed to improving lower extremity muscle power. Squat-to-stand training will stimulate the proprioceptive stimulation on the trunk and lower extremity
  Arms: Lower Limb Fitness Program
Other: Routine Therapy — In control group routine therapy will be given 3 times a week for 6 weeks with session conducting 45 minutes per sessions which involve standing balance exercises, sitting from chair to stand, heal to toe stand will be performed.
  Arms: Routine Therapy

SUMMARY:
Down Syndrome is a congenital disorder resulting from the trisomy of the human chromosome 21, which will determine, among other characteristics, intellectual disability and growth retardation. Reduced muscular strength, cardiovascular capacity, sleep problems, and impaired walking performance are also observed in Down syndrome participants. The estimated global prevalence is around 0.1% of live births. Children with Down's syndrome (DS) often have greater postural sway and delay in motor development. Muscle weakness and hypotonia, particularly of the lower extremities are theorized to impair their overall physical health and ability to perform daily activities. Posture, balance, and movement issues are common in children with Down syndrome. The purpose of this study is to examine the effects of Lower Limb Fitness Program on dynamic balance and mobility in children with Down Syndrome. This study explore that Lower Limb Fitness Program could improve the dynamic balance and mobility in children with DS.

DETAILED DESCRIPTION:
Group A: Experimental group:

Group A will receive Range of motion for 5 minutes involving movements that stretch and strengthen the muscles and improve the stability. Proprioceptive training for 5 minutes which involve Single-leg balance Start with 20-30 seconds per leg and gradually increase to 1 minute 2-3 sets per leg. Weight bearing exercises on an uneven surface (such as Bosu ball or stability disc) and jumping rope 5-10 minutes/session. All proprioceptive training done firstly with eyes open and then with close eyes. Squat-to-stand training proprioceptive training lower extremity. This intervention aims to get the muscles ready before the actual intervention and improve proprioceptive ability. Exercises will be given three times a week for 6 weeks with session conducting 45 minutes per sessions which involve Squat-to-stand training will repeat 30 times 3 sets for 20 min. 2minute break after 1 set.. Balance training which involves standing activities with support, progressing to unsupported as tolerated for 10 minutes/session.

Group B: Control group:

In control group routine therapy will be given 3 times a week for 6 weeks with session conducting 45 minutes per sessions which involve standing balance exercises, sitting from chair to stand, heal to toe stand will be performed.

Data will be assessed by assessor at baseline by single leg stance test and at the end of 6th session of treatment (Pre and post).

ELIGIBILITY:
Inclusion Criteria:

* Age 6-12 years
* Both Genders.
* Single leg stance Test: If unable to stand for 5 seconds or less client at greater risk of injury from fall.
* Ability to understand and follow basic instructions.
* Deficits in Balance

Exclusion Criteria:

* Children who are unable to engage in a structured fitness program due to behavioral or physical limitations.
* Children who have undergone lower limb surgery or experienced significant lower limb injuries in the past six months

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 28 (Actual)
Dates: Start 2024-05-15 (Actual); Primary Completion 2024-07-15 (Actual); Study Completion 2024-07-30 (Actual)

PRIMARY OUTCOMES:
Timed up and go test | 6 weeks
  The TUG test assesses the participant's mobility by timing how quickly they can complete the test and dynamic balance by assessing their ability to sit-to-stand, stand-to-sit, walk, and their ability to change directions. The participant stood up from a chair (46 cm seat height) with no armrests, walked 10 feet, turned around, walked back to the chair, and sat back down as quickly as possible
Pediatric Balance scale | 6 weeks
  Pediatric version of balance scale is used to evaluate static and dynamic balance in children aged 3-15 years with mild-to-moderate motor impairment. The scale comprises 14 items including sitting balance, standing balance, sitting to standing/standing to sitting, transfers, stepping, reaching forward with outstretched arm, retrieving object from floor, turning, and placing foot on stool items. Each item is scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points
Modified Clinical Test of Sensory Interaction in Balance (CTSIB-M) | 6 weeks
  This test is designed to assess how well an older adult is using sensory inputs when one or more sensory systems are compromised. In condition one, all sensory systems (i.e., vision, somatosensory, and vestibular) are available for maintaining balance. In condition two, vision has been removed and the older adult must rely on the somatosensory and vestibular systems to balance

CONTACTS AND LOCATIONS:
Overall Officials: Aqdas Javaid, MS*, Principal Investigator — Riphah International University
Locations (1):
- Riphah International University, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Zai W, Xu N, Wu W, Wang Y, Wang R. Effect of task-oriented training on gross motor function, balance and activities of daily living in children with cerebral palsy: A systematic review and meta-analysis. Medicine (Baltimore). 2022 Nov 4;101(44):e31565. doi: 10.1097/MD.0000000000031565. PMID 36343029